CLINICAL TRIAL: NCT02819908
Title: Dropless™ vs. Less Drops™ Pharmaceutical Regimens After Cataract Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Eye Center of North Florida (Other)
Responsible Party: Principal Investigator, Bret L. Fisher, M.D., Principal Investigator, Eye Center of North Florida
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BF-2015-011
Record Dates: First submitted 2015-09-02; First posted 2016-06-30 (Estimated); Results first posted 2020-03-09 (Actual); Last update posted 2020-03-09 (Actual); Status verified 2020-02

CONDITIONS: Intraocular Lens Associated Postoperative Inflammation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Imprimis Dropless (Active Comparator): TriMoxiVanc 0.2cc intravitreal one time
  Interventions: Drug: Imprimis Dropless
- Imprimis Less Drops (Active Comparator): Pred Moxi, 1 drop tid for 1 week then, PredKeterolac bid for 2-4 weeks.
  Interventions: Drug: Imprimis Less Drops

INTERVENTIONS:
Drug: Imprimis Dropless — Tri-Moxi-Vanc transzonular intravitreal injection
  Arms: Imprimis Dropless
Drug: Imprimis Less Drops — Pred-Moxi-Ketorolac and Pred-Ketorolac topical instillation qd postoperatively
  Arms: Imprimis Less Drops

SUMMARY:
To compare the relative effectiveness of the Imprimis Dropless™ (TriMoxiVanc) intraocular solution with the Less Drops™ topical formulation of PredMoxiKeterolac (given for the first week post op) followed by PredKeterolac (given for weeks 2 to 4 after surgery).

The hypothesis is that the "dropless" regimen will be non-inferior to the "less drops" regimen in terms of post-operative IOP changes, post-operative healing, and visual quality.

DETAILED DESCRIPTION:
Modern cataract surgery has become a relatively short out-patient procedure with small incisions and short post-operative recovery time. Surgery can be influenced by surgical technique and experience. Prophylactic pharmaceutical regimens are designed to control post-operative pain and to reduce the potential for inflammation (i.e. macular edema, CME) and infection (i.e. endophthalmitis).

The most serious potential infection related to cataract surgery is endophthalmitis. Endophthalmitis is a result of microorganisms entering the eye, either during the surgical procedure or before surgical incisions have healed completely. The risk of infection can be reduced in several ways. Pre-operatively, reducing the bacteria on the cornea and ocular adnexa can be helpful. During surgery, appropriate technique can reduce the potential for ingress. Post-operatively, prophylactic antibiotics can eliminate organisms once they have entered the eye. Topical drops, intracameral antibiotics and subconjunctival injections are typical options in current use, usually selected on the basis of spectrum of coverage, cost, efficacy and/or expected side effects.

With regard to inflammation, one of the most common post-operative responses is cystoid macular edema (CME). Steroids and non-steroidal anti-inflammatory drugs (NSAIDs) appear effective in reducing the incidence of CME, with NSAIDs posing a lower risk for IOP spikes and showing greater efficacy some studies.

While there is documented evidence of the utility of prophylactic post-operative treatment for pain and infection, patient compliance remains a significant concern. The regimen is often complex, with multiple drops several times per day. Inability to instill the drops, forgetfulness and a lack of appreciation for the importance of compliance can all be contributing factors.

There are several new options to try to address the potential issues related to poor patient compliance. One is referred to as "dropless" cataract surgery, which involves injection of a multi-drug compound into the eye at time of cataract surgery; one such compound includes triamcinolone acetonide, moxifloxacin hydrochloride and vancomycin (TriMoxiVanc). Another alternative is to reduce the burden of the pharmaceutical regimen using a compounded topical medication; this is termed "less drops" cataract surgery. An option in this regard is a topical formulation of prednisolone acetate, moxifloxacin hydrochloride and ketorolac tromethamine (PredMoxiKetorolac), given for one week post-operatively followed by a topical formulation of prednisolone acetate and ketorolac tromethamine (PredKeterolac) given for weeks 2 to 4 after surgery.

The purpose of this study is to evaluate the differences in performance between the dropless and less-drops pharmaceutical regimens after cataract surgery.

ELIGIBILITY:
Inclusion Criteria:

* Ocular criteria must be met in both eyes.
* Subject is undergoing bilateral cataract extraction or refractive lens exchange with intraocular lens implantation.
* Gender: Males and Females.
* Age: 21 or older.
* Willing and able to provide written informed consent for participation in the study.
* Willing and able to comply with scheduled visits and other study procedures.
* Willing and able to administer eye drops and record the times the drops were instilled.
* Scheduled to undergo standard cataract surgery or refractive lens exchange with topical anesthesia in both eyes within 6-15 days of each other.
* Potential postoperative best-corrected visual acuity of 20/30 or better.

Exclusion Criteria:

* If any of the following exclusion criteria are applicable to the subject or either eye, the subject should not be enrolled in the study.
* Severe preoperative ocular pathology: amblyopia, rubella cataract, proliferative diabetic retinopathy, shallow anterior chamber, macular edema, aniridia or iris atrophy, uveitis, history of iritis, iris neovascularization, medically uncontrolled glaucoma, microphthalmos or macrophthalmos, optic nerve atrophy, macular degeneration (with anticipated best postoperative visual acuity less than 20/30), advanced glaucomatous damage, etc.
* Presence of epiretinal membrane.
* Uncontrolled diabetes.
* Use of any systemic or topical drug known to interfere with visual performance.
* Contact lens use during the active treatment portion of the trial.
* Any concurrent infectious/non-infectious conjunctivitis, keratitis or uveitis.
* History of chronic intraocular inflammation.
* History of retinal detachment.
* Pseudoexfoliation syndrome or any other condition that has the potential to weaken the zonules.
* Previous refractive surgery.
* Anesthesia other than topical, oral or intravenous anesthesia (i.e. retrobulbar, general, etc).
* Any clinically significant, serious or severe medical or psychiatric condition that may increase the risk associated with study participation or may interfere with the interpretation of study results.
* Participation in (or current participation) any investigational drug or device trial within the previous 30 days prior to the start date of this trial.
* Intraocular conventional surgery within the past three months or intraocular laser surgery within one month.

The principal investigator reserves the right to declare a patient ineligible or non-evaluable based on medical evidence that indicates they are unsuitable for the trial.

Exclusion Criteria during surgery:

If any of the following exclusion criteria are applicable to the study eye, the subject should not continue in the study.

* If full dose (0.2 cc) is not delivered into the vitreous through the zonules as evaluated by surgeon's direct visualization of the material in the posterior chamber with lack of material in the anterior chamber and an empty syringe.
* Significant vitreous loss.
* Significant anterior chamber hyphema.
* Uncontrollable intraocular pressure.
* Zonular or capsular rupture.
* Bag-sulcus, sulcus-sulcus or unknown placement of the haptics.
* Suturing of incision required at time of surgery.
* Intraocular lens tilt or decentration
* Peri-bulbar or retro-bulbar block required during surgery.
* Other procedure, such as pupil stretch, expanders, iris hooks during surgery.

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2015-09; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bret L Fisher, MD, Principal Investigator — Eye Center of North Florida
Locations (1):
- Eye Center of North Florida, Panama City, Florida, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Imprimis Dropless | Imprimis Less Drops
Started (25 patients total of 50 eyes) | 12 | 13
Completed | 12 | 13
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Study data has been lost to natural disaster (Hurricane Micheal), therefore there is no study data that is available to report
Groups:
- Total: Total of all reporting groups
Arm/Group | Imprimis Dropless | Imprimis Less Drops | Total
Number analyzed (Participants) | 0 | 0 | 0
Age, Categorical
Age, Continuous
Sex: Female, Male
Region of Enrollment [unit: participants]

OUTCOME MEASURES:

1. Primary Outcome: The Change in Intraocular Pressure (IOP) From Baseline
Description: Based on Goldmann tonometry
Time Frame: To end of study (1 month postop)
Population: as for baseline characteristics
Groups:
- Imprimis Dropless: TriMoxiVanc 0.2cc intravitreal one time
  Imprimis Dropless: Tri-Moxi-Vanc transzonular intravitreal injection
  no Adverse events
- Imprimis Less Drops: Pred Moxi, 1 drop tid for 1 week then, PredKeterolac bid for 2-4 weeks.
  Imprimis Less Drops: Pred-Moxi-Ketorolac and Pred-Ketorolac topical instillation qd postoperatively
  No adverse events
Arm/Group | Imprimis Dropless | Imprimis Less Drops
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Change in Corneal Thickness
Description: Based on corneal pachymetry
Time Frame: To end of study (1 month postop)
Population: as for baseline characteristics
Arm/Group | Imprimis Dropless | Imprimis Less Drops
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Slit Lamp (Cornea Exam)
Time Frame: To end of study (1 month postop)
Population: as for baseline characteristics
Arm/Group | Imprimis Dropless | Imprimis Less Drops
Number analyzed (Participants) | 0 | 0

4. Other Pre Specified Outcome: Subject Reporting no Eye Pain
Description: "0"( on the eye pain/discomfort scale)
Time Frame: To end of study (1 month postop)
Population: as for baseline characteristics
Arm/Group | Imprimis Dropless | Imprimis Less Drops
Number analyzed (Participants) | 0 | 0

5. Other Pre Specified Outcome: Change From Baseline Eye Pain/Discomfort
Description: eye pain/discomfort scale
Time Frame: To end of study (1 month postop)
Population: as for baseline characteristics
Arm/Group | Imprimis Dropless | Imprimis Less Drops
Number analyzed (Participants) | 0 | 0

6. Other Pre Specified Outcome: The Proportion of Subjects Reporting no Visual Symptoms ("0" )
Description: visual symptom scale
Time Frame: To end of study (1 month postop)
Population: as for baseline characteristics
Arm/Group | Imprimis Dropless | Imprimis Less Drops
Number analyzed (Participants) | 0 | 0

7. Other Pre Specified Outcome: The Change From Baseline in Visual Symptoms
Description: visual symptom scale
Time Frame: To end of study (1 month postop)
Population: as for baseline characteristics
Arm/Group | Imprimis Dropless | Imprimis Less Drops
Number analyzed (Participants) | 0 | 0

8. Other Pre Specified Outcome: The Change From Baseline in Central Corneal Thickness Measurements
Description: corneal pachymetry
Time Frame: To end of study (1 month postop)
Population: as for baseline characteristics
Arm/Group | Imprimis Dropless | Imprimis Less Drops
Number analyzed (Participants) | 0 | 0

9. Other Pre Specified Outcome: The Change From Baseline in Macular Thickness Measurements
Description: based on optical coherence tomography (OCT) measurement
Time Frame: To end of study (1 month postop)
Population: as for baseline characteristics
Arm/Group | Imprimis Dropless | Imprimis Less Drops
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Study data has been lost to natural disaster (Hurricane Micheal), therefore there is no study data that is available to report
Description: Study data has been lost to natural disaster (Hurricane Micheal), therefore there is no study data that is available to report
Arm/Group | Imprimis Dropless | Imprimis Less Drops
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
Study data has been lost to natural disaster (Hurricane Micheal), therefore there is no study data that is available to report

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No